CLINICAL TRIAL: NCT02727803
Title: Personalized NK Cell Therapy in CBT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0313; NCI-2016-00584 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0313 (Other: M D Anderson Cancer Center); R01CA211044 (NIH)
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Acute Myeloid Leukemia With Variant MLL Translocations; B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Chemotherapy-Related Leukemia; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; ISS Stage II Plasma Cell Myeloma; ISS Stage III Plasma Cell Myeloma; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts; Myelodysplastic Syndrome With Gene Mutation; Myelodysplastic/Myeloproliferative Neoplasm; Previously Treated Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Refractory Acute Lymphoblastic Leukemia; Refractory Adult Acute Lymphoblastic Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Antilymphocyte Serum; Busulfan; Clofarabine; Cyclophosphamide; fludarabine phosphate; Melphalan; Rituximab; CT-P10; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Myeloablative regimen 1 (Experimental): Patients receive anti-thymocyte globulin IV over 4 hours on days -9 and -8, fludarabine phosphate IV over 1 hour, clofarabine IV over 1 hour, and busulfan IV over 3 hours on days -7 to -4. Patients undergo TBI on day -3.
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo umbilical cord blood transplantation on day 0.
  NK CELLS INFUSION: Patients receive NK cells IV over 30 minutes between days 30-180.
  Interventions: Biological: Allogeneic Natural Killer Cell Line NK-92; Biological: Anti-Thymocyte Globulin; Drug: Busulfan; Drug: Clofarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation
- Non-myeloablative regimen 2 (Experimental): Patients with CD20 positive malignancies receive rituximab IV over 6 hours on day -9. Patients receive anti-thymocyte globulin IV over 4 hours on days -8 and -7, fludarabine phosphate IV over 1 hour on days -6 to -3, and cyclophosphamide IV over 3 hours on day -6 and undergo TBI on day -1 at the discretion of the investigator(s).
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo umbilical cord blood transplantation on day 0.
  NK CELLS INFUSION: Patients receive NK cells IV over 30 minutes between days 30-180.
  Interventions: Biological: Allogeneic Natural Killer Cell Line NK-92; Biological: Anti-Thymocyte Globulin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Rituximab; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation
- Reduced intensity regimen 3 (Experimental): Patients receive anti-thymocyte globulin IV over 4 hours on days -7 and -6, fludarabine phosphate IV over 1 hour on days -5 to -2, and melphalan IV over 30 minutes on day -2.
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo umbilical cord blood transplantation on day 0.
  NK CELLS INFUSION: Patients receive NK cells IV over 30 minutes between days 30-180.
  Interventions: Biological: Allogeneic Natural Killer Cell Line NK-92; Biological: Anti-Thymocyte Globulin; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Biological: Allogeneic Natural Killer Cell Line NK-92 — Given IV
  Other Names: haNK; NK-92; NK-92 Cells
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATS
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
  Arms: Myeloablative regimen 1
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
  Arms: Myeloablative regimen 1
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Non-myeloablative regimen 2
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Reduced intensity regimen 3
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
  Arms: Non-myeloablative regimen 2
Radiation: Total-Body Irradiation — Undergo total body irradiation
  Other Names: Total Body Irradiation; Whole-Body Irradiation
  Arms: Myeloablative regimen 1; Non-myeloablative regimen 2
Procedure: Umbilical Cord Blood Transplantation — Undergo umbilical cord blood transplantation
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This phase II clinical trial studies how well personalized natural killer (NK) cell therapy works after chemotherapy and umbilical cord blood transplant in treating patients with myelodysplastic syndrome, leukemia, lymphoma or multiple myeloma. This clinical trial will test cord blood (CB) selection for human leukocyte antigen (HLA)-C1/x recipients based on HLA-killer-cell immunoglobulin-like receptor (KIR) typing, and adoptive therapy with CB-derived NK cells for HLA-C2/C2 patients. Natural killer cells may kill tumor cells that remain in the body after chemotherapy treatment and lessen the risk of graft versus host disease after cord blood transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression-free survival (PFS) time.

SECONDARY OBJECTIVES:

I. Overall survival (OS) time. II. Transplant related mortality (TRM). III. Graft versus host disease (GVHD). IV. Infection

OUTLINE: Patients are assigned to 1 of 3 preparative regimens.

MYELOABLATIVE REGIMEN 1: Patients receive anti-thymocyte globulin intravenously (IV) over 4 hours on days -9 and -8, fludarabine phosphate IV over 1 hour, clofarabine IV over 1 hour, and busulfan IV over 3 hours on days -7 to -4. Patients undergo total body irradiation (TBI) on day -3.

NON-MYELOABLATIVE REGIMEN 2: Patients with cluster of differentiation (CD)20 positive malignancies receive rituximab IV over 6 hours on day -9. Patients receive anti-thymocyte globulin IV over 4 hours on days -8 and -7, fludarabine phosphate IV over 1 hour on days -6 to -3, and cyclophosphamide IV over 3 hours on day -6 and undergo TBI on day -1 at the discretion of the investigator(s).

REDUCED INTENSITY REGIMEN 3: Patients receive anti-thymocyte globulin IV over 4 hours on days -7 and -6, fludarabine phosphate IV over 1 hour on days -5 to -2, and melphalan IV over 30 minutes on day -2.

UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo umbilical cord blood transplantation on day 0.

NK CELLS INFUSION: Patients receive NK cells IV over 30 minutes between days 30-180.

After completion of study treatment, patients are followed up at 1, 7, 14, 28, 45, 60, and 100 days, and at 6, 9, and 12 months, and then yearly for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following hematologic malignancies: acute myelogenous leukemia (AML), induction failure, high-risk for relapse first remission (with intermediate-risk or high-risk cytogenetics including complex karyotype, abnormal [abn][3q], -5/5q-, -7/7q-, abn[12p], abn[17p], myeloid/lymphoid or mixed-lineage leukemia [MLL] gene re-arrangement and t [6;9]47, fms related tyrosine kinase 3 [flt3] mutation positive and/or evidence of minimal residual disease by flow cytometry), secondary leukemia from prior chemotherapy and/or arising from myelodysplastic syndromes (MDS), any disease beyond first remission
* Myelodysplastic syndrome (MDS): Primary or therapy related, including patients that will be considered for transplant; these include any of the following categories: 1) revised International Prognostic Scoring System (IPSS) intermediate and high risk groups, 2) malondialdehyde (MDA) with transfusion dependency, 3) failure to respond or progression of disease on hypomethylating agents, 4) refractory anemia with excess of blasts, 5) transformation to acute leukemia, 6) chronic myelomonocytic leukemia, 7) atypical MDS/myeloproliferative syndromes, 8) complex karyotype, abn(3g), -5/5g-, -7/7g-, abn(12p), abn(17p)
* Acute lymphoblastic leukemia (ALL): Induction failure, primary refractory to treatment (do not achieve complete remission after first course of therapy) or are beyond first remission including second or greater remission or active disease; patients in first remission are eligible if they are considered high risk, defined as any of the following detected at any time: with translocations 9;22 or 4;11, hypodiploidy, complex karyotype, secondary leukemia developing after cytotoxic drug exposure, and/or evidence of minimal residual disease or acute biphenotypic leukemia, or double hit non-Hodgkin's lymphoma
* Non-Hodgkin's lymphoma (NHL) in second or third complete remission, or relapse (including relapse post autologous hematopoietic stem cell transplant); relapsed double hit lymphomas; patients with options for treatment that are known to be curative are not eligible
* Small lymphocytic lymphoma (SLL), or chronic lymphocytic leukemia (CLL) with progressive disease following a minimum of two lines of standard therapy
* Chronic myeloid leukemia (CML) second chronic phase or accelerated phase
* Hodgkin's disease (HD): Induction failures, after first complete remission, or relapse (including relapse post autologous hematopoietic stem cell transplant), or those with active disease
* Multiple myeloma: stage II or III, symptomatic, secretory multiple myeloma requiring treatment
* A person (such as a haploidentical family member) or unit of cord blood must be identified as a source of back-up cells source in case of engraftment failure
* Patient age criteria: age >= 15 and =< 45 years (myeloablative regimen 1; age >= 15 and =< 80 years (nonmyeloablative regimen 2) at the discretion of the investigator(s); age >= 15 and =< 80 years old that in the opinion of the investigator(s) would preclude myeloablative therapy may receive reduced intensity regimen 3
* Performance score of at least 60% by Karnofsky
* Left ventricular ejection fraction of at least 40% (myeloablative regimen 1, reduced intensity regimen 3)
* Left ventricular ejection fraction of at least 30% (nonmyeloablative regimen 2)
* Pulmonary function test (PFT) demonstrating an adjusted diffusion capacity of least 50% predicted value for hemoglobin concentration (myeloablative regimen 1, reduced intensity regimen 3)
* Serum creatinine within normal range, or if serum creatinine outside normal range, then renal function (measured or estimated creatinine clearance or glomerular filtration rate [GFR]) > 40mL/min/1.73 m^2
* Serum glutamate pyruvate transaminase (SGPT)/bilirubin < to 2.0 x normal (myeloablative regimen 1), reduced intensity regimen 3; SGPT/bilirubin < to 4.0 x normal (nonmyeloablative regimen 2)
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months
* Patients with options for treatment that are known to be curative are not eligible
* Patients enrolled in this study may be enrolled on other supportive care investigational new drug (IND) studies at the discretion of the principal investigator (PI)

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive; HIV results will be determined by nucleic acid testing
* Uncontrolled serious medical condition such as persistent septicemia despite adequate antibiotic therapy, decompensated congestive heart failure despite cardiac medications or pulmonary insufficiency requiring intubation (excluding primary disease for which cord blood [CB] transplantation is proposed), or psychiatric condition that would limit informed consent
* Active central nervous system (CNS) disease in patient with history of CNS malignancy
* Availability of appropriate, willing, human leukocyte antigen (HLA)-matched related stem cell donor

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) time in C2C2 patients | From the date of engraftment to disease progression or death, assessed up to 4 years
  Distributions of time-to-event variables will be estimated using the method of Kaplan and Meier, and Bayesian regression models will be used to assess the relationship of each outcome with patient covariates, including disease stage, KIR haplotype, age, diagnosis, human leukocyte antigen (HLA) match, cytomegalovirus (CMV) status, and gender. Categorical outcomes will be evaluated by tabulation and Bayesian regression modeling.
Progression free survival (PFS) time in C1 patients | From the date of cord blood transplant to disease progression or death, assessed up to 4 years
  Distributions of time-to-event variables will be estimated using the method of Kaplan and Meier, and Bayesian regression models will be used to assess the relationship of each outcome with patient covariates, including disease stage, KIR haplotype, age, diagnosis, HLA match, CMV status, and gender. Categorical outcomes will be evaluated by tabulation and Bayesian regression modeling.

SECONDARY OUTCOMES:
Overall survival time | Up to 4 years
  Distributions of time-to-event variables will be estimated using the method of Kaplan and Meier, and Bayesian regression models will be used to assess the relationship of each outcome with patient covariates, including disease stage, KIR haplotype, age, diagnosis, HLA match, CMV status, and gender. Categorical outcomes will be evaluated by tabulation and Bayesian regression modeling.
Incidence of transplant related mortality | Up to 4 years
  Bayesian regression models will be used to assess the relationship of each outcome with patient covariates, including disease stage, KIR haplotype, age, diagnosis, HLA match, CMV status, and gender. Categorical outcomes will be evaluated by tabulation and Bayesian regression modeling.
Incidence of graft-versus host disease | Up to 4 years
  Bayesian regression models will be used to assess the relationship of each outcome with patient covariates, including disease stage, KIR haplotype, age, diagnosis, HLA match, CMV status, and gender. Categorical outcomes will be evaluated by tabulation and Bayesian regression modeling.
Incidence of infection | Up to 4 years
  Bayesian regression models will be used to assess the relationship of each outcome with patient covariates, including disease stage, KIR haplotype, age, diagnosis, HLA match, CMV status, and gender. Categorical outcomes will be evaluated by tabulation and Bayesian regression modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Olson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org